CLINICAL TRIAL: NCT00177203
Title: Agewise Project 3: Brief Behavioral Treatment of Insomnia in Primary Care
Acronym: AW3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 021115; 5P01AG020677 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Insomnia
Keywords: Insomnia; Sleep Disorders; Sleeplessness; Chronic Insomnia; Sleep Studies; Disorders of Initiating and Maintaining Sleep; Primary Care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment of Insomnia or Information — The behavioral treatment involves education about sleep and its disorders; habits that help and hurt sleep; and recommendations about sleep hours and time in bed. It involves two meetings with a nurse who is part of the research team.
  In the information condition, participants are given similar information in printed brochures that are published by the American Academy of Sleep Medicine. They are instructed to read the information.
  Other Names: Information only

SUMMARY:
This project will test the efficacy of a brief, 2 session behavioral intervention for insomnia, as compared to an information-only condition. We hypothesize that compared to those receiving the information-only intervention, those assigned to BBTI will have superior short-term outcomes and retain the gains made, at 12 months.

We will also compare older insomniacs to age matched good sleepers through measurers of mental and physical health, sleep, and general functioning. We hypothesize that the insomnia cohort will have more physical and mental health disorders of a greater severity than the age-matched controls.

DETAILED DESCRIPTION:
As a prevalent problem among the elderly, insomnia is often treated by primary care physicians, and benzodiazepine receptor agonists (BzRA) are the most widely prescribed form of treatment. Behavioral interventions offer an effective option to BzRA therapy as they are preferred by many elderly patients and have a lower side effect profile. Presently behavioral interventions are available on specialty care clinics, provided by trained therapists, requiring up to six intervention sessions. This project will test the efficacy of a brief, two sessions behavioral model which could be adapted to the primary care setting. In addition, we will compare older insomniacs to age matched good sleepers through measurers of mental and physical health, sleep and general functioning. We expect that 100 enrolled individuals age 60 or older with Insomnia and a control cohort of 50 enrolled individuals matched by age and gender will complete the study. Subjects will be randomly assigned to one of two intervention conditions: (1.) receive a two session Brief Behavioral Treatment Intervention(BBTI), or (2.) a information-only modality in which they will be encouraged to read handouts on sleep, insomnia and healthy sleep practices published by the AASM. Clinical evaluation will include the Agebat measures (common to all five projects in this Program Project) and in-home or laboratory polysomnographic measures. Sleep dairies and wrist actigraphy will be used to measure treatment adherence. Patients will be evaluated before and after completing the assigned intervention cells. Those receiving BBTI will be re-evaluated at 12 months following a six month "booster" session. Data obtained from the control cohort will include the Agebat measures. We hypothesize that compared to those receiving the information-only intervention, those assigned to BBTI will have superior short-term outcomes and retain the gains made, at 12 months. We also predict that the insomnia cohort will have more physical and mental health disorders of a greater severity than the age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Current diagnosis of Insomnia using DSM-IV criteria (Insomnia group)
* No current diagnosis of Insomnia (Control group)
* Provision of written informed consent

Exclusion Criteria:

* Psychiatric: untreated depressive, anxiety, psychotic and substance use disorders and/or treated or untreated delirium of dementia. We will exclude at intake to the study any individual with moderate to severe cognitive impairment who is likely to be demented. In the event that an individual scores less than < 25 on the Mini-Mental State Exam, we will exclude that person from the study. We will also discuss our concerns with the subject and will suggest that he or she contact the Memory Disorders Clinic run by the Alzheimer's Disease Research Center. We will give the subject literature on this Clinic as well as their phone number. We will not exclude persons with milder cognitive decrements because chronic medical disease and its associated sleep disruption are themselves associated with some impairment of cognitive performance.
* Medical: ongoing chemotherapy or radiation cancer treatment, hospitalization within the past two weeks or terminal illness with a life expectancy less than 6 months;
* Sleep: untreated obstructive sleep apnea syndrome, narcolepsy or restless legs syndrome.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Short-term outcome will be assessed by administration of the AgeWise battery of assessments (Agebat) and polysomnographic evaluations pre and post intervention. | Short-term outcome is assessed 4 weeks after intervention begins.
Durability of BBTI will be evaluated by readministration of the clinical portions of the Agebat at six months, and both the clinical and polysomnographic evaluations at twelve months. | 6 months and 12 months after the start of the intervention

SECONDARY OUTCOMES:
We will evaluate the effects of physical and mental health on sleep during the initial evaluation. We will also determine how physical and mental health affects response to the specific sleep interventions at week 4, and 6 and 12 months. | Week 4, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Buysse, M.D., Principal Investigator — University of Pittsburgh Medical Center, Western Psychiatric Institute & Clinic
Locations (1):
- University of Pittsburgh Medical Center, Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Buysse DJ, Germain A, Moul DE, Franzen PL, Brar LK, Fletcher ME, Begley A, Houck PR, Mazumdar S, Reynolds CF 3rd, Monk TH. Efficacy of brief behavioral treatment for chronic insomnia in older adults. Arch Intern Med. 2011 May 23;171(10):887-95. doi: 10.1001/archinternmed.2010.535. Epub 2011 Jan 24. PMID 21263078